CLINICAL TRIAL: NCT02126618
Title: The Effect of Diuresis During 20-minute Pad Test on the Estimation of the Severity of Stress Urinary Incontinence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201403054RIND
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower urinary tract symptoms; urodynamic studies; diuresis
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- women with lower urinary tract symptoms

SUMMARY:
The aim of this study is to estimate the amount of extra urine produced by natural diuresis during 20-minute pad test, and assess the effect of diuresis on the accuracy of using 20-minute pad test to estimate the severity of SUI. Besides, the above results may be used for further refinement of the amount of water infusion used for the 20-minute pad test.

DETAILED DESCRIPTION:
Pad testing is an important method to evaluate the severity of women with stress urinary incontinence (SUI). The investigators had proved the superiority of the infusion of the strong desire amount while using 20-minute pad test for detecting SUI. However, a considerable volume of urine may be produced by natural diuresis during the course of 20-minute pad test with strong-desire amount infusion, and may cause bladder overdistension, more urine leakage and overestimate the severity of SUI. Thus, the aim of this study is to estimate of the amount of extra urine produced by natural diuresis, and assess its effect on the ability of using pad weight to estimate the severity of SUI.

The investigators will review the clinical data of patients who receiving urodynamic studies in the Department of Obstetrics & Gynecology of National Taiwan University Hospital between January 2008 and March 2014. STATA 11.0 software will be used for statistical analysis.

The investigators will get the mean values of diuresis, and the factors affecting the amount of diuresis. Besides, the investigators can get the influence of diuresis on the accuracy of 20-minute pad test as a role of estimating the severity of SUI. The above data should be important for further refinement of 20-minute pad test.

ELIGIBILITY:
Inclusion Criteria:

* More than 20-year-old woman who with stress urinary incontinence (SUI).
* We will review the clinical data, urodynamics, pad weight and bladder diary of patients who receiving urodynamic studies and 20-minute pad test in the Department of Obstetrics & Gynecology of National Taiwan University Hospital between January 2008 and March 2014.

Exclusion Criteria:

* < 20 year old female

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with lower urinary tract symptoms and underwent urodynamic testing
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Estimation of natural diuresis during pad testing | 7 years
  The aim of this study is to estimate the amount of extra urine produced by natural diuresis, and assess its effect on the ability of using pad weight to estimate the severity of SUI.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics & Gynecology, National Taiwan University Hospital, Taipei, Taiwan